CLINICAL TRIAL: NCT02056119
Title: Randomized Controlled Trial of Mesh Versus Jet Nebulizers on Clinical Outcomes During Mechanical Ventilation in the Intensive Care Unit
Brief Title: RCT of Mesh Versus Jet Nebulizers on Clinical Outcomes During Mechanical Ventilation in the Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 13070203
Record Dates: First submitted 2014-01-15; First posted 2014-02-05 (Estimated); Results first posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Respiratory Insufficiency
Keywords: Ventilators, mechanical; Aerosol Drug Therapy; Nebulizers; Equipment Contamination; vibrating mesh nebulizer; jet nebulizer; mechanical ventilation; ventilator associated event; ventilator associated tracheobronchitis
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Jet Nebulizer Arm (Active Comparator): The Jet Nebulizer Protocol:
  * Physician order received for subject, randomization to jet nebulizer occurred.
  * Jet nebulizer, Misty Max 10™ (Carefusion, CA), placed into spring loaded t-piece between the humidifier and the ventilator (approximately 15 cm from the gas outlet).
  * Aerosol treatment delivered per physician order at flow rates of 8-10 L/min.
  * Jet nebulizer to be replaced every 3 days per hospital protocol. a. Prior to every nebulizer change or every 3 days, study staff to be notified in order to obtain cultures.
  Interventions: Device: Jet Nebulizer Arm
- Vibrating Mesh Nebulizer Arm (Experimental): * Physician order received for subject, randomization to vibrating mesh nebulizer occurred.
  * Aeroneb® Solo (Aerogen, Galway, Ireland) vibrating mesh nebulizer to be placed before the heater on the "dry side" of the heater water chamber on the inspiratory ventilator circuit.
  * Aerosol treatment delivered per physician order.
  * Mesh nebulizer to be replaced every 30 days per hospital protocol. a. Prior to every nebulizer change or every 3 days, study staff to be notified in order to obtain cultures.
  Interventions: Device: Vibrating Mesh Nebulizer Arm

INTERVENTIONS:
Device: Vibrating Mesh Nebulizer Arm — * Physician order received for subject, randomization to vibrating mesh nebulizer occurred.
  * Aeroneb® Solo (Aerogen, Galway, Ireland) vibrating mesh nebulizer to be placed before the heater on the "dry side" of the heater water chamber on the inspiratory ventilator circuit.
  * Aerosol treatment delivered per physician order.
  * Mesh nebulizer to be replaced every 30 days per hospital protocol. a. Prior to every nebulizer change or every 3 days, study staff to be notified in order to obtain cultures.
  Other Names: Aeroneb Solo (Aerogen, Galway, Ireland)
  Arms: Vibrating Mesh Nebulizer Arm
Device: Jet Nebulizer Arm — * Physician order received for subject, randomization to jet nebulizer occurred.
  * Jet nebulizer, Misty Max 10™ (Carefusion, CA), placed into spring loaded t-piece between the humidifier and the ventilator (approximately 15 cm from the gas outlet).
  * Aerosol treatment delivered per physician order at flow rates of 8-10 L/min.
  * Jet nebulizer to be replaced every 3 days per hospital protocol. a. Prior to every nebulizer change or every 3 days, study staff to be notified in order to obtain cultures.
  Other Names: Misty Max 10 nebulizer (Carefusion, California)
  Arms: Jet Nebulizer Arm

SUMMARY:
Aerosol delivery during mechanical ventilation has long been a long debated topic. As evidence-based knowledge about the delivery of aerosol to the lungs of mechanically ventilated patients increases, one piece of the puzzle has remained unexplored; measurement of clinically relevant outcomes. The primary aim of this research is to compare clinical outcomes (ventilator-associated events (VAEs), length of stay (LOS) in intensive care unit (ICU), and total days on mechanical ventilation) when using a traditional jet nebulizer versus a newer generation vibrating mesh nebulizer during mechanical ventilation. The secondary aim of this research is to identify source of bacteria by obtaining cultures of each nebulizer and ventilator circuit and plating them for colony growth and identification.

DETAILED DESCRIPTION:
This pilot study was designed as a randomized, controlled trial comparing clinical outcomes and contamination rates in jet nebulizers versus vibrating mesh nebulizers. The sample size will be one of consecutive convenience over an entire year (September 2013-September 2014) to include all seasons. The study will be performed at Rush University Medical Center (RUMC) in Chicago, IL.

Each mechanically ventilated patient within inclusion criteria, with a physician order for aerosol treatment, will be randomized to either the jet nebulizer or mesh nebulizer group using SPSS computer software. The respiratory care staff will place the nebulization device in the ventilator circuit per hospital protocol. Both devices, jet and mesh nebulizers, are currently standard practice; therefore hospital protocol will be followed regarding placement and administration of ordered aerosol treatment.

The study subject will remain on the device to which they were randomized for the duration of their hospital stay to obtain clinical outcome data. Study staff to be notified of patient extubation from mechanical ventilation, discharge from intensive care unit, or expiration; this will conclude participant involvement in the study. Retrospective clinical outcome data will be obtained from the subject's electronic medical chart at conclusion of study.

Retrospective data to include:

1. LOS in ICU (days)
2. LOS on mechanical ventilator (days)
3. Drug administration information

   1. Drug and dose ordered
   2. Number of treatments delivered
   3. Treatment type

      * Continuous
      * Intermittent
4. Ventilator-Associated Tracheobronchitis (# VATs)16

   a. Fever, increased volume and purulence of secretions, a positive culture (quantitative or semi-quantitative) of a respiratory sample (tracheal aspirates or bronchoscopic specimens), and the absence of a new or an evolving pulmonary infiltrate in the chest x-ray in a patient on mechanical ventilation >48 hours
5. Ventilator-Associated Events in Adults15

   1. Ventilator-Associated Condition (# VACs)

      * After a period of stability or improvement on the ventilator, the patient has at least one of the following indications of worsening oxygenation:
      * Minimum daily FiO2 values increase ≥ 0.20 over baseline and remain at or above that increased level for ≥ 2 calendar days. -
      * Minimum daily PEEP values increase ≥ 3 cm H2O over baseline and remain at or above that increased level for ≥ 2 calendar days.
   2. Infection-related Ventilator-Associated Complication (# IVACs)

      * On or after calendar day 3 of mechanical ventilation and within 2 calendar days before or after the onset of worsening oxygenation, the patient meets both of the following criteria:
      * Temperature > 38˚ C or < 36˚ C, or white blood cell count ≥ 12,000 cells/mm3 or ≤ 4,000 cells/mm3. AND
      * A new antimicrobial agent(s) is started, and is continued for ≥ 4 calendar days.
   3. Possible Ventilator-Associated Pneumonia (# Possible VAPs)

      * On or after calendar day 3 of mechanical ventilation and within 2 calendar days before or after the onset of worsening oxygenation, ONE of the following criteria is met:
      * Purulent respiratory secretions
      * Positive culture
   4. Probably Ventilator-Associated Pneumonia (# Probable VAPs)

      * On or after calendar day 3 of mechanical ventilation and within 2 calendar days before or after the onset of worsening oxygenation, ONE of the following criteria is met:
      * Purulent respiratory secretions (from one or more specimen collections- and defined as for possible VAP) and one of the following (positive culture of endotracheal aspirate, positive culture of bronchoalveolar lavage, positive culture of lung tissue, positive culture of protected specimen brush
      * One of the following without requirement for purulent respiratory secretions (positive pleural fluid culture, positive lung histopathology, positive diagnostic test for Legionella, positive diagnostic test on respiratory secretions for influenza virus, respiratory syncytial virus, adenovirus, parainfluenza virus)

The Jet Nebulizer Protocol:

* Physician order received for subject; randomization to jet nebulizer occurred.
* Jet nebulizer, Misty Max 10™ (Carefusion, CA), placed into spring-loaded t-piece between the humidifier and the ventilator (approximately 15 cm from the gas outlet).
* Aerosol treatment delivered per physician order at flow rates of 8-10 L/min.
* Jet nebulizer to be replaced every 3 days per hospital protocol.

  1. Prior to every nebulizer change or every 3 days, study staff to be notified in order to obtain cultures.
  2. Cultures

     * Jet Nebulizer Culture (3 plates): Sample to be collected from jet nebulizer by running oxygen at a flow of 8-10 L/min through nebulizer (3 mL normal saline in the reservoir) while directing the nebulizer towards plate for 1 minute. Process to be repeated for 3 different plates. Plates to be labeled, have edges sealed with tape, be placed in biohazard bag and sent to microbiology lab for analysis.

       1. Plate 1: MacConkey agar (id gram (-) organisms)
       2. Plate 2: Chocolate agar (id fastidious organisms)
       3. Plate 3: Blood agar (id gram(+) and gram(-) organisms)
     * Ventilator Circuit Culture: Material to be collected from rim of inspiratory ventilator circuit at wye by rubbing a sterile swab along circuit 3x in a circular motion. Swab to be sealed in test tube with lid and sent to lab for analysis.
     * Sputum samples: Data obtained per electronic medical chart. Sputum sample data to be analyzed in study when ordered by physician.
* After obtaining cultures, the jet nebulizer will be replaced with new one and labeled per hospital protocol.
* Further cultures are not necessary unless patient is identified by study staff to have VAE. (Appendix A)
* Study staff to be notified of patient extubation from mechanical ventilation, discharge from intensive care unit or expiration.

The Vibrating Mesh Nebulizer protocol:

* Physician order received for subject; randomization to vibrating mesh nebulizer occurred.
* Aeroneb® Solo (Aerogen, Galway, Ireland) vibrating mesh nebulizer to be placed before the heater on the "dry side" of the heater water chamber on the inspiratory ventilator circuit.
* Aerosol treatment delivered per physician order.
* Mesh nebulizer to be replaced every 30 days per hospital protocol.

  1. Prior to every nebulizer change or every 3 days, study staff to be notified in order to obtain cultures.
  2. Cultures

     * Vibrating Mesh Nebulizer Culture (3 plates): Sample to be collected from vibrating mesh nebulizer while directing the nebulizer(3 mL normal saline in the reservoir) towards plate for 1 minute. Process to be repeated for 3 different plates. Plates to be labeled, have edges sealed with tape, be placed in biohazard bag and sent to microbiology lab for analysis.

       1. Plate 1: MacConkey agar (id gram (-) organisms)
       2. Plate 2: Chocolate agar (id fastidious organisms)
       3. Plate 3: Blood agar (id gram(+) and gram(-) organisms)
     * Ventilator Circuit Culture: Material to be collected from rim of inspiratory ventilator circuit at wye by rubbing a sterile swab along circuit 3x in a circular motion. Swab to be sealed in test tube with lid and sent to lab for analysis.
     * Sputum samples: Data obtained per electronic medical chart. Sputum sample data to be analyzed in study when ordered by physician.
* Vibrating mesh nebulizer replaced with new one and labeled per hospital protocol.
* Further cultures not necessary unless patient identified by study staff to have VAE. (appendix A)
* Study staff to be notified immediately of patient extubation from mechanical ventilation, discharge from intensive care unit or expiration.

ELIGIBILITY:
Inclusion Criteria:

* Age > 1 y/o
* Intubated with endotracheal tube (ETT) and on mechanical ventilation
* Patient in all intensive care units at Rush University Medical Center
* Physician order for aerosolized breathing treatment in medical record

Exclusion Criteria:

* Age < 1 y/o
* Diaphragmatic paralysis
* Paraplegic or high spinal cord injury
* Brain death

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-09; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meagan N Dubosky, MS, Principal Investigator — Rush University, Respiratory Care Research Coordinator
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The sample size was one of consecutive convenience (September 2013- August 2014). This study included adult subjects, greater than 18 years of age, receiving mechanical ventilation through an endotracheal tube (ETT) in the intensive care unit (ICU) with a physician order for aerosol treatment. Excluded were subjects receiving mechanical ventilation through a tracheostomy or diagnosed with diaphragmatic paralysis, paraplegia, high spinal cord injury, or brain death.
Groups:
- Jet Nebulizer Arm: The Jet Nebulizer Protocol:
  * Physician order received for subject, randomization to jet nebulizer occurred.
  * Jet nebulizer, Misty Max 10™ (Carefusion, CA), placed into spring loaded t-piece between the humidifier and the ventilator (approximately 15 cm from the gas outlet).
  * Aerosol treatment delivered per physician order at flow rates of 8-10 L/min.
  * Jet nebulizer to be replaced every 3 days per hospital protocol. a. Prior to every nebulizer change or every 3 days, study staff to be notified in order to obtain cultures.
  Jet Nebulizer Arm: •Physician order received for subject, randomization to jet nebulizer occurred.
  * Jet nebulizer, Misty Max 10™ (Carefusion, CA), placed into spring loaded t-piece between the humidifier and the ventilator (approximately 15 cm from the gas outlet).
  * Aerosol treatment delivered per physician order at flow rates of 8-10 L/min.
  * Jet nebulizer to be replaced every 3 days per hospital protocol. a. Prior to every nebulizer change or every
- Vibrating Mesh Nebulizer Arm: * Physician order received for subject, randomization to vibrating mesh nebulizer occurred.
  * Aeroneb® Solo (Aerogen, Galway, Ireland) vibrating mesh nebulizer to be placed before the heater on the "dry side" of the heater water chamber on the inspiratory ventilator circuit.
  * Aerosol treatment delivered per physician order.
  * Mesh nebulizer to be replaced every 30 days per hospital protocol. a. Prior to every nebulizer change or every 3 days, study staff to be notified in order to obtain cultures.
  Vibrating Mesh Nebulizer Arm: •Physician order received for subject, randomization to vibrating mesh nebulizer occurred.
  * Aeroneb® Solo (Aerogen, Galway, Ireland) vibrating mesh nebulizer to be placed before the heater on the "dry side" of the heater water chamber on the inspiratory ventilator circuit.
  * Aerosol treatment delivered per physician order.
  * Mesh nebulizer to be replaced every 30 days per hospital protocol. a. Prior to every nebulizer change or every 3 days, study staf
Period: Overall Study
Arm/Group | Jet Nebulizer Arm | Vibrating Mesh Nebulizer Arm
Started | 58 | 62
Completed | 48 | 42
Not Completed | 10 | 20
Not completed — Death | 1 | 2
Not completed — Intubated for less than 24 hrs | 2 | 7
Not completed — No aerosol treatments were given. | 3 | 2
Not completed — Received Metaneb treatment | 0 | 2
Not completed — Protocol Violation | 4 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Jet Nebulizer Arm | Vibrating Mesh Nebulizer Arm | Total
Number analyzed (Participants) | 48 | 42 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.5 (16.2) | 64.0 (13.8) | 62.1 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 21 | 43
  Male | 26 | 21 | 47
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black | 20 | 9 | 29
  Race: White | 17 | 22 | 39
  Race: Hispanic | 3 | 5 | 8
  Race: Asian | 3 | 0 | 3
  Race: Indian | 0 | 1 | 1
  Race: Other | 4 | 3 | 7
  Race: Unknown | 1 | 2 | 3
The Acute Physiology and Chronic Health Evaluation (APACHE II) [Mean (Standard Deviation); unit: units on a scale] — This score ranges from 0 to 71. The higher the score the more the patient's illness is.
  units on a scale | 20.6 (7.6) | 21.3 (8.6) | 20.9 (8.0)

OUTCOME MEASURES:

1. Primary Outcome: Venilator Associated Events (VAE)
Description: Ventilator associated conditions (VAC) and infection related ventilator associated conditions (IVAC) were identified based on the 2013 NHSN Surveillance for VAEs (e,g., "See page 92 at https://www.cdc.gov/nhsn/PDFs/pscManual/validation/2013-PSC-Manual-validate.pdf for detailed criteria.")
Time Frame: duration of mechanical ventilation or discharge from the intensive care unit
Measure: Count of Participants; unit: Participants
Groups:
- Jet Nebulizer Arm: The Jet Nebulizer Protocol:
  * Physician order received for subject, randomization to jet nebulizer occurred.
  * Jet nebulizer, Misty Max 10™ (Carefusion, CA), placed into spring loaded t-piece between the humidifier and the ventilator (approximately 15 cm from the gas outlet).
  * Aerosol treatment delivered per physician order at flow rates of 8-10 L/min.
  * Jet nebulizer to be replaced every 3 days per hospital protocol. a. Prior to every nebulizer change or every 3 days, study staff to be notified in order to obtain cultures.
  Jet Nebulizer Arm: •Physician order received for subject, randomization to jet nebulizer occurred.
  * Jet nebulizer, Misty Max 10™ (Carefusion, CA), placed into spring loaded t-piece between the humidifier and the ventilator (approximately 15 cm from the gas outlet).
  * Aerosol treatment delivered per physician order at flow rates of 8-10 L/min.
  * Jet nebulizer to be replaced every 3 days per hospital protocol. a. Prior to every nebulizer change or every 3 days, study staff to be notified in order to obtain cultures.
- Vibrating Mesh Nebulizer Arm: * Physician order received for subject, randomization to vibrating mesh nebulizer occurred.
  * Aeroneb® Solo (Aerogen, Galway, Ireland) vibrating mesh nebulizer to be placed before the heater on the "dry side" of the heater water chamber on the inspiratory ventilator circuit.
  * Aerosol treatment delivered per physician order.
  * Mesh nebulizer to be replaced every 30 days per hospital protocol. a. Prior to every nebulizer change or every 3 days, study staff to be notified in order to obtain cultures.
  Vibrating Mesh Nebulizer Arm: •Physician order received for subject, randomization to vibrating mesh nebulizer occurred.
  * Aeroneb® Solo (Aerogen, Galway, Ireland) vibrating mesh nebulizer to be placed before the heater on the "dry side" of the heater water chamber on the inspiratory ventilator circuit.
  * Aerosol treatment delivered per physician order.
  * Mesh nebulizer to be replaced every 30 days per hospital protocol. a. Prior to every nebulizer change or every 3 days, study staff to be notified in order to obtain cultures.
Arm/Group | Jet Nebulizer Arm | Vibrating Mesh Nebulizer Arm
Number analyzed (Participants) | 48 | 42
Participants
  Ventilator Associated Conditions: No | 44 | 40
  Ventilator Associated Conditions: Yes | 4 | 2
  Infection Related Ventilator Associated Conditions: No | 46 | 42
  Infection Related Ventilator Associated Conditions: Yes | 2 | 0

2. Secondary Outcome: Participants With Bacterial Growth
Description: While on mechanical ventilator, bacterial growth will be assessed from the vent circuit and nebulizer, and participant sputum.
Time Frame: duration of mechanical ventilation or discharge from the intensive care unit
Population: Cultures were not obtained for all participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Jet Nebulizer Arm | Vibrating Mesh Nebulizer Arm
Number analyzed (Participants) | 47 | 42
Participants
  Growth in Nebulizer: No | 41 | 30
  Growth in Nebulizer: Yes | 6 | 12
  Growth in Circuit: number analyzed (Participants) | 44 | 42
  Growth in Circuit: No | 26 | 13
  Growth in Circuit: Yes | 18 | 29
  Growth in Sputum Culture: number analyzed (Participants) | 21 | 23
  Growth in Sputum Culture: No | 7 | 3
  Growth in Sputum Culture: Yes | 14 | 20

3. Secondary Outcome: Length of Stay in Intensive Care Unit
Description: Total length of stay in intensive care unit in days
Time Frame: discharge from the intensive care unit
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Jet Nebulizer Arm | Vibrating Mesh Nebulizer Arm
Number analyzed (Participants) | 48 | 42
Days | 11.0 (8.3) | 14.1 (11.8)

4. Secondary Outcome: Days on Mechanical Ventilation
Description: Total days spent on Mechanical Ventilator
Time Frame: discharge from the intensive care unit
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Jet Nebulizer Arm | Vibrating Mesh Nebulizer Arm
Number analyzed (Participants) | 48 | 42
Days | 6.7 (7.1) | 9.7 (9.4)

ADVERSE EVENTS:
Time Frame: Adverse events were collected through study completion, an average of 14 days.
Arm/Group | Jet Nebulizer Arm | Vibrating Mesh Nebulizer Arm
All-Cause Mortality (participants affected / at risk) | 14/48 | 15/42
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/42
Other Adverse Events (participants affected / at risk) | 0/48 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes